CLINICAL TRIAL: NCT06506682
Title: Blinded, Randomized Trial Comparing Constraint Induced Movement Therapy With Virtual Reality to Constraint Induced Movement Therapy Alone and the Correlation of Patient Characteristics With Responsiveness to Intervention
Brief Title: Comparing CIMT With Virtual Reality to CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 2021-0271
Record Dates: First submitted 2024-05-29; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT (Active Comparator): Both groups will participate in 60 hours of intensive therapy over 10 days at SRC (6 hours per day Monday-Friday) following the established 'Pirate Camp' CIMT protocol. The full protocol can be found at: https://twu.edu/occupational-therapy/Camp-Based-Augmented-CIMT-Guide/. Both groups will participate in child friendly outdoor and indoor activities that promote the use of the involved side for example; parachute games, sock toss, penny pick up.
  Interventions: Behavioral: Constraint Induced Movement Therapy
- CIMT+VR (Experimental): The CIMT+VR group will use the VR technology to work on upper limb motor skills for approximately two hours per day (4 of the activities described under Key Information at the beginning of this form) while the CIMT-only group will participate in traditional motor-based task-specific activities. Both the VR games and traditional intervention will target the improvement of the same upper limb domains.
  Interventions: Behavioral: CIMT + VR

INTERVENTIONS:
Behavioral: Constraint Induced Movement Therapy — CIMT is an intensive upper limb therapy for children with unilateral (one sided) cerebral palsy where the child wears a constraint (splint or mit) on their dominant hand so that they use the involved (weaker) side to do activities
  Other Names: CIMT
  Arms: CIMT
Behavioral: CIMT + VR — Participants in the CIMT+VR group of this study protocol will do everything the CIMT group does PLUS will utilize at least 4 of the following VR technologies each day of intervention: FitMi, Tyromotion Pablo® UpperExtremity, Hocoma Armeo® Spring Pediatric, Nintendo Wii, and Parrot Drone.
  Arms: CIMT+VR

SUMMARY:
This study is being done to compare constraint induced movement therapy (CIMT) to CIMT combined with virtual reality technology (CIMT+VR) and its impact on how the children with unilateral cerebral palsy use their arm. CIMT is an intensive upper limb therapy for children with one sided (unilateral) cerebral palsy where the child wears a constraint (splint or mit) on their dominant hand so that they use the involved (weaker) side to do activities. Both groups will work on using both arms together to complete activities (bimanual training) as a way to transfer newly learned skills with one hand into two handed tasks. Assessments before and after the intervention will include clinical assessments (where a research team member observes the child doing tasks and ask questions), motion capture (where the child's movement is recorded using multiple cameras), and wearable sensors on the wrists (like a watch).

DETAILED DESCRIPTION:
The purpose of this research study is to compare the effectiveness of constraint induced movement therapy (CIMT) to CIMT combined with virtual reality technology (CIMT+VR) in children with unilateral cerebral palsy. Both groups will also work on bimanual training (using both arms together to complete activities) as a way to transfer newly learned skills with one hand into two handed tasks. One group will receive CIMT, and the other group will receive CIMT and the VR technology. CIMT is an intensive upper limb therapy for children with unilateral (one sided) cerebral palsy where the child wears a constraint (splint or mit) on their dominant hand so that they use the involved (weaker) side to do activities. Participants in the CIMT+VR group of this study protocol will do everything the CIMT group does PLUS will utilize at least 4 of the following VR technologies each day of intervention: FitMi, Tyromotion Pablo Upper Extremity, Hocoma Armeo® Spring Pediatric, Nintendo Wii, and Parrot Drone.

FitMi is a neurorehabilitation device that provides visual feedback on motor performance as the individual interacts with wireless switches (Flint Rehab, 2020). The targeted areas of upper limb function for the study include grasp, release, and thumb opposition.

Tyromotion Pablo® Upper Extremity is a sensor based rehabilitation device with interactive therapies for the whole body. It provides targeted training for pronation/supination and force regulation for gross grasp, tip pinch, lateral and three point pinch (Tyromotion). The targeted areas of upper limb function for the study include supination, grip strength, and pinch strength.

Hocoma Armeo® Spring Pediatric is a device that combines the assistance of an exoskeleton and VR games created to improve hand function in the pediatric population. The Hocoma Armeo ® Spring Pediatric encourages repetitive movement of the UL with the aim of increasing quantity and improving quality of movements and can be customized for range of motion and the amount of gravity assistance the exoskeleton provides the child while playing the VR games. The targeted areas of upper limb function for the study include upper arm movement and wrist extension.

Nintendo Wii® is a video game console that uses a handheld pointing device that detects movement in three directions. The system requires the individual to hold the controller in the hand while moving the upper extremity. The targeted areas of upper limb function for the study include stabilize and hold. Parrot Drone is a stable quadcopter mini drone that can be flown indoors and outdoors. It has an autopilot feature that keeps the drone steady even if the user lets go of the controller. The drone can be controlled with a remote control or from a smart device that will target isolated finger and thumb movements.

Participants may exit the study prior to completion of the program due to non-compliance, social and economic barriers, disease progression, misdiagnosis or no longer meeting inclusion criteria. Caregivers may withdraw their child from the study at any time for any reason.

Participants enrolled in the study will complete (1) baseline assessments, including physical assessments with motion capture, which will require a visit to Scottish Rite for Children (SRC), (2) an upper limb intervention program that will require visits to Scottish Rite each weekday for two weeks, and (3) post-intervention assessments, including physical assessments with motion capture, that will require a visit to Scottish Rite, for a total of 12 visits. Assessment visits will each take about 3 hours and group intervention sessions will last 6 hours each day. Participants will also be asked as an option to wear an accelerometer (ActiGraph) on their wrists during waking hours (approximately 12 hours per day) 2-3 days before and after the intervention and during the 2 weeks of intervention for a total of 16-18 days. Total study duration for participants will be about 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* have cerebral palsy (a brain injury that causes muscle movement problems) or are a non-progressive brain injury to the developing brain and have difficulty using one of your arms

Exclusion Criteria:

* unable to complete assessment protocol

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | Baseline, pre-intervention and immediate post-intervention
  assessment of bimanual hand skills in children with cerebral palsy well the involved hand performs during two handed activities,

SECONDARY OUTCOMES:
Melbourne Unilateral Upper Limb Assessment (MUUL) | Baseline, pre-intervention and immediate post-intervention
  how well the involved hand works and active range of motion
ICF Brief Core Set for Cerebral Palsy | Baseline, pre-intervention
  Interview based on ICR Core Set
Hypertonia Assessment Tool Assessment Tool (HAT) | Baseline, pre-intervention and immediate post-intervention
  tone assessment
Canadian Occupational Performance Measure Occupational Performance Measure (COPM) | Baseline, pre-intervention and immediate post-intervention
  Goal setting
sensory assessment | Baseline, pre-intervention and immediate post-intervention
  assess sensory of hand stereognosis, two point discrimination, proprioception,
motion capture with electromyography (EMG) | Baseline, pre-intervention and immediate post-intervention
  while completing the AHA
option wearing of ActiGraphs on upper limbs | Baseline, pre-intervention and immediate post-intervention
  real time tracking of use of upper extremities

CONTACTS AND LOCATIONS:
Locations (1):
- Scottish Rite for Children, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No